CLINICAL TRIAL: NCT04007965
Title: Novel Technique of Pneumatic Posterior Capsulorhexis for Treatment and Prevention of Posterior Capsular Opacification
Acronym: PCO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Shaaban Elwan, Assistant professor of ophthalmology, Minia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Minia University
Record Dates: First submitted 2019-06-29; First posted 2019-07-05 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Posterior Capsule Opacification
Keywords: PCO

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Opacified posterior capsule (Experimental): PCO
  Interventions: Procedure: Pneumatic Posterior Capsulorhexis
- Clear posterior capsule (Active Comparator): CPC
  Interventions: Procedure: Pneumatic Posterior Capsulorhexis

INTERVENTIONS:
Procedure: Pneumatic Posterior Capsulorhexis — Pneumatic Posterior Capsulorhexis using air dose 0.1 ml and Healon dose 0.5 -1.0 ml.

SUMMARY:
ABSTRACT PURPOSE: To evaluate a new technique of posterior capsulorhexis using air support to treat primary posterior capsular opacification (PCO) during cataract extraction surgery or to prevent post-operative PCO.

SETTING: 1-Ophthalmology department, Faculty of medicine, Minia University, El-Minia, Egypt.

2- Security Forces Hospital, Ophthalmology Department, Riyadh, Kingdom of Saudi Arabia.

DESIGN: Prospective, randomized case-control comparative study.

Methods: 100 eyes of 100 patients with a mean age of 63.3 years with dens cataract. Fifty of them ( group 1) with primary PCO (discovered during the operations) and fifty (group 2) with clear posterior capsule.

All cases undergone phacoemulsification, posterior capsulorhexis using the air to support the posterior capsule and separate it from the vitreous (the novel technique will be discussed later). Then IOL implantations wear done in the bag between the anterior and posterior capsular rim. Each patient was evaluated for the following:- visual acuity (UCVA and BCVA), intraocular pressure, intra ocular lens stability, visual axis opacification and posterior segment complications as retinal break, retinal detachment or cystoid macular oedema.

DETAILED DESCRIPTION:
Introduction. Posterior capsular opacification (PCO) is one of the common late post-operative complications of phacoemulsification and ECCE. The treatment of PCO by YAG laser capsulotomy usually leads to the famous annoying symptom (musca) and carries the risk of IOP elevation. Moreover, it may lead to the posterior segment complications ( cystoid macular edema, retinal breaks and detachment). There is no reliable treatment for prevention of PCO.

The current available modalities to prevent postoperative PCO are:

* Some surgical modifications as hydrodissection, repeated nucleus rotation and meticulous polishing of the lens epithelial cells (LECs) from anterior capsular rim and equator. In 1989 David Apple and his group (1) had demonstrated the value of hydrodissection. In 1992, they further emphasized hydrodissection as well as barriers to migration of equatorial cells to the posterior capsule as methods which could reduce PCO (2). In the same year Fine described a technique which he termed 'cortical cleaving hydrodissection', (3) which was designed to break the equatorial adhesions between lens epithelial cells and the capsule, thus increasing the chance of significant clearance of these cells which are the progenitors of PCO. In 2006 they pointed out to the laboratory and clinical evidence that good hydrodissection, coupled with mechanical 'scouring' of LECs from the equator may have beneficial effect on decreasing PCO incidence. (4,5). In a laboratory experiment they found that there were significantly fewer cells remaining in the capsule equator in the group of eyes where the lens had been rotated three times within the bag prior to removal, compared with no such rotation(4).
* Changes in the IOL design and materials: e.g. The square edge of the optic and acrylic IOL decreases the incidence of postoperative PCO than with PMMA IOLs of similar design.
* Pharmacological strategies either to kill the residual epithelial cells or to prevent their post operative proliferation. The pharmacological prevention has been largely unsuccessful so far. Moreover, any agent must be toxic to these epithelial cells without being toxic to the corneal endothelium. Few agents have been partially successful without clinical application till now (6).

The incidence of PCO following successful cataract surgery has been falling since the general acceptance of posterior chamber in-the-bag intraocular lens (IOL) implantation. Improvement in lens materials, lens design and technique are well documented to decrease the incidence of postoperative PCO (8, 9). Rotation three times of the hydrodissected nucleus prior to phacoemulsification and a second hydrodissection after nucleus removal are simple and safe maneuvers that statistically improve the results (9). Bimanual irrigation/aspiration may also help.(10) Treatment options for PCO

* YAG laser posterior capsulotomy
* Surgical posterior capsulotomy or capsulectomy
* Primary (Intra-operative)
* Secondary.

Patients and methods:

Indications of the new technique

1. Intraoperative PCO in white cataract.
2. As a primary procedure during cataract extraction to prevent post-operative PCO. Thirty eyes of 100 patients with dens cataract were chosen from the outpatient clinic of the ophthalmology department, Minia University Hospital, El-Minia Egypt. The patient's age ranged from 50-73 years with a mean age of 63.3 years 50 males and 50 females without any local or systemic causes for the cataract. The study group included fifty eyes (group1) with PCO, and fifty eyes (group 2) with clear posterior capsule (discovered intra-operative). All cases were subjected to complete ophthalmic examinations and echographic data registration. All cases undergone Phacoemulsification, posterior capsulorhexis using the air to support the posterior capsule and separate it from the vitreous face. Table (1)

The novel technique:

After complete phacoemulsification of the nucleus and I/A:

1. Visco-elastic material was injected to make the anterior chamber formed without deepening so that the posterior capsule is not forcibly pushed backward.
2. The posterior capsule punctured centrally using cysteotome Fig. (1).
3. Controllable one shot injection of 0.1 ml of sterile air through the posterior capsule puncture which elevate, support and separate the posterior capsule from vitreous face. (Insulin syringe and Helon cannula were used) Fig. (2).
4. Another visco-elastic injection to the anterior chamber to stretch the posterior capsule and sandwitich it between visco-elastic above and the air below Fig. (3).
5. Posterior capsulorhexis 4-5 mm is now performed easily using capsulorhexis forceps then foldable IOL was implanted between the anterior and posterior capsular rim .

ELIGIBILITY:
Inclusion Criteria:

* Dense mature cataract without any local or systemic causes for the cataract.

Exclusion Criteria:

* Any patients did not complete the follow up visits
* younger patients and children

Ages: 50 Years to 73 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2019-06-25 (Actual)

PRIMARY OUTCOMES:
Visual acuity measured using snellen chart projector | one year
  visual acuity (UCVA and BCVA) measured in decimal values
IOP measured in numerical values | one year
  Intra-ocular pressure measured by Tono pen
IOL stability | one year
  Intraocular Lens stability seen by slit lamb examination
Visual Axis Opacification | 0ne year
  Visual Axis Opacification seen by slit lamb examination

SECONDARY OUTCOMES:
posterior segment complications | 18 months
  posterior segment complications as retinal break, retinal detachment or cystoid macular oedema.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Eid, MD, Study Chair — Minia University
Locations (1):
- Security forces hospital, Riyadh, Central, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Walker TD. Pharmacological attempts to reduce posterior capsule opacification after cataract surgery--a review. Clin Exp Ophthalmol. 2008 Dec;36(9):883-90. doi: 10.1111/j.1442-9071.2009.01921.x. PMID 19278485
- [Derived] Eid AM, Abd-Elhamid Mehany Elwan S, Sabry AM, Moharram HM, Bakhsh AM. Novel Technique of Pneumatic Posterior Capsulorhexis for Treatment and Prevention of Posterior Capsular Opacification. J Ophthalmol. 2019 Dec 21;2019:3174709. doi: 10.1155/2019/3174709. eCollection 2019. PMID 31949950